CLINICAL TRIAL: NCT03209479
Title: Copaxone Subcutaneous Injection Syringe Special Drug Use-Result Investigation (All-Case Investigation) "Prevention of Relapse of Multiple Sclerosis"
Status: Completed | Type: Observational
Sponsor: Teva Takeda Pharma Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: Glatiramer-5001; jRCT1080223004 (Registry Identifier: jRCT)
Record Dates: First submitted 2017-07-04; First posted 2017-07-06 (Actual); Last update posted 2024-06-13 (Actual); Status verified 2024-06

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis | interventions — Glatiramer Acetate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Glatiramer acetate: For adults, a 20 mg dose of glatiramer acetate will be subcutaneously administered once daily. Participants will receive interventions as part of routine medical care.
  Interventions: Drug: Glatiramer acetate

INTERVENTIONS:
Drug: Glatiramer acetate — Copaxone subcutaneous injection syringe
  Other Names: Copaxone subcutaneous injection syringe

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of Copaxone subcutaneous injection syringe (hereinafter referred to as Copaxone) in patients with multiple sclerosis in the routine clinical setting.

DETAILED DESCRIPTION:
The drug being tested in this study is called Glatiramer acetate is being tested to treat people who have Multiple sclerosis. This study will look at the safety and efficacy of Glatiramer acetate in patients with multiple sclerosis in the routine clinical setting.

The study will enroll approximately 1000 patients.

• Glatiramer acetate subcutaneous injection syringe

This multi-center trial will be conducted in Japan.

ELIGIBILITY:
Inclusion Criteria:

- All patients treated with Copaxone from the first day of market launch of the product

Exclusion Criteria:

-None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population will consist of all participants with a diagnosis of multiple sclerosis and received their first dose of Copaxone/glatiramer acetate.
Sampling Method: Probability Sample
Enrollment: 1332 (Actual)
Dates: Start 2015-11-24 (Actual); Primary Completion 2024-03-31 (Actual); Study Completion 2024-03-31 (Actual)

PRIMARY OUTCOMES:
Percentage of participants who had one or more adverse events | Up to 24 months
Annual Relapse Rate (ARR) | Up to 24 months
  The annual relapse rate (ARR) after the start of treatment will be calculated throughout study.

SECONDARY OUTCOMES:
Changes in the number of lesions from brain MRI findings | Up to 24 months
Changes in functional evaluation scores (Expanded Disability Status Scale [EDSS]) | Up to 24 months
  EDSS is a method of quantifying disability in multiple sclerosis and monitoring changes in the level of disability over time. EDSS scale ranges from 0 to 10 in 0.5 unit increments and higher score refers to people with higher levels of disability by multiple sclerosis.
Changes in functional evaluation scores (Functional Systems [FS]) | Up to 24 months
  FS is based on a standard neurological examination; the 7 functional systems plus "other" (Pyramidal, Cerebellar, Brainstem, Sensory, Bowel and bladder function, Visual function, Cerebral [or mental] functions, other) are rated. Each FS is scored on a scale of 0 (no disability) to 5 or 6 (more severe disability), and total score ranging from 0 to 40. Higher score in each functional system refers to people with higher levels of disability by multiple sclerosis.

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda (Note: This product was divested to Teva Takeda Pharma Ltd. in 2024.)
Locations (1):
- Takeda selected site, Tokyo, Japan

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.

REFERENCES:
- See also: To obtain more information on the study, click here/on this link — https://clinicaltrials.takeda.com/study-detail/5f6b60234db2bf003ab49722